CLINICAL TRIAL: NCT03957070
Title: The Sonic Incytes Liver Incyte System, Assessment of Liver Fibrosis and Steatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonic Incytes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SI-CLIN-01
Record Dates: First submitted 2019-04-03; First posted 2019-05-21 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Liver Fibrosis; Liver Steatosis
Keywords: liver; ultrasound elastography
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Liver Incyte (Experimental): Patients with successfully treated HCV, or NASH Healthy volunteers with no history of liver disease. Patients and Volunteers will be scanned with FibroScan and Liver Incyte.
  Interventions: Device: Liver Incyte

INTERVENTIONS:
Device: Liver Incyte — Ultrasound elasticity imaging

SUMMARY:
Evaluate the feasibility of the Liver Incyte system for liver elasticity measurement in healthy volunteers and patients with liver fibrosis. To evaluate the discriminatory ability of elasticity measurements generated by Liver Incyte for healthy volunteers versus patients with liver fibrosis in comparison to FibroScan measurements.

DETAILED DESCRIPTION:
This will be a prospective, open label, feasibility and validation study of the Liver Incyte system in patients with liver fibrosis (Cohort 1, n = 150) and healthy volunteers (Cohort 2, n = 50), for a total of 200 participants. The physician operator of the FibroScan, and the operator of the Shear wave vibro-elastography (S-WAVE) system, will not be blinded to the clinical diagnoses of the patients. All patients will undergo the testing with both FibroScan and Liver Incyte system at a single in-clinic visit.

The liver stiffness of each participant will be assessed with the Liver Incyte Model B device and with FibroScan. The elasticity measurements from these two devices will be the primary outcome measure.

The Liver Incyte system is designed as two models with differences in the ultrasound components only, description of the two models is below. Two sub-studies are included in this design as exploratory objectives. Model B will be utilized at all study sites and all study participants. Participants at the LAIR study site will also be evaluated using Model A, as well as Model B, for verification and to confirm consistency between designs. Participants will have the option to participate in the Magnetic Resonance Elastography (MRE) and Proton Density Fat Fraction (PDFF) portion of the study. MRE/PDFF is an optional procedure, which makes up a sub-study for this trial, this would require approximately 1 hour, and is open to any participant who is willing and has time for the extra study visit. The results of the MRE/PDFF sub-study will be included as an exploratory objective.

ELIGIBILITY:
Inclusion Criteria:

* Any sex, ages 19-75 years inclusively
* Individuals with a history of chronic Hepatitis C (HCV) or non-alcoholic steatohepatitis (NASH). Patients with history of Hepatitis C must have completed treatment and achieved Sustained viral response at 12 weeks (SVR12).
* Previous FibroScan measurement (within the last 13 months) between 8 kilopascals and 35 kilopascals.
* Able to understand the informed consent form, study procedures and willing to participate in study

Exclusion Criteria:

* Unable to achieve SVR12 with previous antiviral treatment for HCV
* Multiple (>1) liver disease diagnoses within the past 12 months
* Co-infection with another Hepatitis virus or Human Immunodeficiency Virus (HIV), last testing within past 5 years
* Documented or known ascites
* Documented or known portal hypertension
* BMI greater than 35 kg/m2 (30 kg/m2 for optional MRE participants)
* If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
* Individuals with history of persistent ethanol abuse (alcohol consumption exceeding 2 standard drinks per day on average [1 standard drink = 10 grams of alcohol])
* Individuals with implanted electrical devices such as pacemakers, internal defibrillators, cochlear implants and nerve stimulators.
* Individuals with surgically removed gallbladder (for optional MRE procedure only)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Discrimination of healthy from patients with liver fibrosis | 6 months
  The discriminatory ability of elasticity measurements generated by Liver Incyte for healthy volunteers versus patients with liver fibrosis in comparison to FibroScan measurements.
  An receiver operating characteristic (ROC) curve using final Liver Incyte elasticity measurement as a predictor of healthy versus fibrotic (HCV/NASH) will be constructed with accompanying 95% confidence interval for the area under the curve (AUC). The AUC and 95% confidence intervals for the FibroScan device will be calculated.

SECONDARY OUTCOMES:
Safety of the device as measured by rate of adverse events | 6 months
  The safety and tolerability of the Liver Incyte system for liver elasticity measurement in healthy volunteers and patients with liver fibrosis
  Rate of adverse events when using the investigational device will be reported.

OTHER OUTCOMES:
Agreement between Liver Incytes and MRI elastography measurements | 6 months
  Elasticity measurements from Liver Incyte and MRE will be compared using a concordance correlation coefficient and associated 95% confidence intervals. A Spearman correlation coefficient and 95% confidence intervals will also be calculated. As in the analysis for the Primary Objective, an ROC curve will be constructed and AUCs for differentiating healthy versus fibrotic (HVC/NASH) will be calculated.
Correlation between Liver Incytes and MRI elastography measurements | 6 months
  Steatosis measurements from Liver Incyte, Fibroscan (CAP), and MRI (PDFF) will be compared using a concordance correlation coefficient and associated 95% confidence intervals. A Spearman correlation coefficient and 95% confidence intervals will also be calculated. An ROC curve will be constructed and AUCs for differentiating healthy versus fibrotic (HCV/NASH) will be calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States
- LAIR, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curry MP, Tam E, Schneider C, Abdelgelil N, Hassanien T, Afdhal NH. The Use of Noninvasive Velacur(R) for Discriminating between Volunteers and Patients with Chronic Liver Disease: A Feasibility Study. Int J Hepatol. 2024 Jan 17;2024:8877130. doi: 10.1155/2024/8877130. eCollection 2024. PMID 38274398